CLINICAL TRIAL: NCT03374891
Title: DECIDE - ICD: A Multicenter Trial of a Shared DECision Support Intervention for Patients Offered Implantable Cardioverter-DEfibrillators
Brief Title: A Multicenter Trial of a Shared DECision Support Intervention for Patients Offered Implantable Cardioverter-DEfibrillators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-1697; 1R01HL136403-01 (NIH)
Record Dates: First submitted 2017-11-29; First posted 2017-12-15 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Systolic; Heart Failure
Keywords: Shared Decision Making;; Defibrillator
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: Step-wedge design. 6 groups will begin recruiting participants as control participants. Throughout the study, at 5 month intervals, 1 randomly selected site at a time will begin intervention.
  Due to the impact of COVID-19 on sites and patient visits from March-April 2020, we moved back the implementation of intervention dates for the 5th site (UCH/DH) by 2 months and the 6th site (Beth Israel) by 1 month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants will fill out surveys (No Intervention): These participants will fill out surveys in regard to their experiences, opinions, and knowledge of the defibrillator process.
- Educational video and/or handout (Active Comparator): These participants will receive an educational video and/or handout about the defibrillator process. Then they will fill out surveys in regard to their experiences, opinions, and knowledge of the defibrillator process.
  Interventions: Other: Educational video and/or handout

INTERVENTIONS:
Other: Educational video and/or handout — The intervention includes a video and/or handout (whichever is easier for the participant) that will give information about defibrillators and about other patients' experiences with their decisions about defibrillators.
  Arms: Educational video and/or handout

SUMMARY:
The investigators goal is to assess real-world effectiveness of patient decision aids (PtDA) for high-risk decisions using the implantable cardioverter-defibrillator (ICD) as a model.

DETAILED DESCRIPTION:
The investigators propose the DECIDE-ICD trial: a type II effectiveness implementation hybrid trial of the investigators ICD PtDAs. The Investigators will use a 6-site stepped-wedge design, with implementation guided by normalization process theory® and evaluation guided by the RE-AIM framework.

The investigators aim to evaluate reach and effectiveness of the ICD PtDAs using a pragmatic, stepped-wedge design on decision quality (knowledge and value-concordance) and psychosocial outcomes.

* Hypothesis 1a: PtDAs will reach over 50% of eligible patients.
* Hypothesis 1b: ICD PtDAs will be effective in improving decision quality in real-world practice.
* Hypothesis 1c: Better informed patients will have lower anxiety, higher rates of planning for the possibility of deactivation, and increased identification of a surrogate decision maker.

The investigators propose 3 a priori hypotheses:

* The decision aids will have a differential effect on the decisions of participants by age (>= 70 years old vs <70 years old);
* The decision aids will have a differential effect on the decisions of participants by heart failure type (non-ischemic vs ischemic);
* The decision aids will have a differential effect on the decisions of participants by the type of device they are considering (ICD vs ICD replacement vs CRT-D).

Along with these hypotheses, we recognize that other important covariates exist, such as health literacy and education level.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking (videos and surveys have only been validated in English)
* Patients have been offered a primary prevention ICD for initial implant, reimplantation, or CRT with defibrillation

Exclusion Criteria:

* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Matlock, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Knoepke CE, Wallace BC, Allen LA, Lewis CL, Gupta SK, Peterson PN, Kramer DB, Brancato SC, Varosy PD, Mandrola JM, Tzou WS, Matlock DD. Experiences Implementing a Suite of Decision Aids for Implantable Cardioverter Defibrillators: Qualitative Insights From the DECIDE-ICD Trial. Circ Cardiovasc Qual Outcomes. 2022 Nov;15(11):e009352. doi: 10.1161/CIRCOUTCOMES.122.009352. Epub 2022 Nov 15. PMID 36378770

RESULTS

PARTICIPANT FLOW:
Groups:
- Surveys Only: These participants will fill out surveys in regard to their experiences, opinions, and knowledge of the defibrillator process.
- Educational Video and/or Handout + Surveys: These participants will receive an educational video and/or handout about the defibrillator process. Then they will fill out surveys in regard to their experiences, opinions, and knowledge of the defibrillator process.
  Educational video and/or handout: The intervention includes a video and/or handout (whichever is easier for the participant) that will give information about defibrillators and about other patients' experiences with their decisions about defibrillators.
Period: Overall Study
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys
Started | 346 | 444
Completed | 323 | 437
Not Completed | 23 | 7

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only collected for participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys | Total
Number analyzed (Participants) | 323 | 437 | 760
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66 [56 to 73] | 67 [58 to 74] | 66.5 [56 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 120 | 209
  Male | 234 | 317 | 551
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 18 | 42
  Not Hispanic or Latino | 299 | 419 | 718
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 5 | 13
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 47 | 84
  White | 250 | 339 | 589
  More than one race | 10 | 16 | 26
  Unknown or Not Reported | 16 | 28 | 44
Region of Enrollment [Number; unit: participants]
  United States | 323 | 437 | 760

OUTCOME MEASURES:

1. Primary Outcome: Knowledge About Defibrillation at Baseline
Description: Multiple survey responses by participants will indicate knowledge changes over time. The Decision Quality Knowledge Survey measures knowledge about defibrillators. Possible scores range from 0 to 100, with higher scores indicating more knowledge and better outcomes.
Time Frame: Baseline
Population: Data was not able to be collected for all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys
Number analyzed (Participants) | 312 | 412
score on a scale | 53.4 (17.6) | 55.4 (17.0)

2. Primary Outcome: Knowledge About Defibrillation at 1 Month
Description: as for outcome 1
Time Frame: 1 month
Population: Data was not able to be collected for all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys
Number analyzed (Participants) | 253 | 370
score on a scale | 57.1 (18.2) | 58.0 (15.4)

3. Primary Outcome: Knowledge About Defibrillation at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: Data was not able to be collected for all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys
Number analyzed (Participants) | 245 | 343
score on a scale | 56.6 (17.4) | 58.6 (14.5)

4. Secondary Outcome: Reach of Eligible Patients
Description: Measuring how many patients of the eligible patient base are able to view or read the educational materials.
Time Frame: Baseline
Population: The control group did not receive the intervention, and was not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys
Number analyzed (Participants) | 0 | 437
Participants
  Were administered intervention by hospital |  | 349
  Were not administered intervention by hospital |  | 88

5. Other Pre Specified Outcome: Differential Effect by Age
Description: The decision aids will have a differential effect on the decisions of participants by age (>= 70 years old vs <70 years old)
Time Frame: Baseline, 1 month, 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Differential Effect by Heart Failure Type
Description: The decision aids will have a differential effect on the decisions of participants by heart failure type (non-ischemic vs ischemic)
Time Frame: Baseline, 1 month, 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Differential Effect by Type of Device
Description: The decision aids will have a differential effect on the decisions of participants by the type of device they are considering (ICD vs ICD replacement vs CRT-D).
Time Frame: Baseline, 1 month, 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Serious Adverse Events and All cause Mortality were not collected for this study for any participant, due to the design of this implementation study. The only participants that were at risk for the incomplete consent process adverse event were the participants enrolled at the one site which required a separate written HIPAA authorization.
Arm/Group | Surveys Only | Educational Video and/or Handout + Surveys
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/346 | 0/444
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Surveys Only (N=346) | Educational Video and/or Handout + Surveys (N=444)
Incomplete consent process (Investigations) | 3/9 (3) | 0/51 (0) — Participants consented verbally, which was not an complete consent process due to HIPAA written consent requirements. HIPAA waiver later obtained. Only participants enrolled at 1 site with separate written HIPAA authorization were at risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03374891/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03374891/ICF_001.pdf